CLINICAL TRIAL: NCT03774199
Title: NightOwl Pulse Oximeter Calibration Study
Acronym: NPOCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ectosense NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-023U1.1
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Pulse Oximeter Calibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulse oximeter calibration population (Other)
  Interventions: Device: NightOwl

INTERVENTIONS:
Device: NightOwl — The NightOwl is a finger and/or forehead mounted device with, among other functions, the capability to acquire double-wavelength PPG, from which SpO2 can be derived

SUMMARY:
Calibration of a software module that computes SpO2 based on photoplethysmography (PPG) traces acquired by a reflectance-based pulse oximeter which can be placed on the index finger or the forehead.

The study is designed in accordance with Medical electrical equipment - Part 2-61: Particular requirements for basic safety and essential performance of pulse oximeter equipment (ISO 80601- 2-61:2011)

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects (ASA 1 and ASA 2) upon signing the informed consent. (ASA : american society of anesthesiologist's health score)

Exclusion Criteria:

* smokers or individuals exposed to high levels of carbon monoxide that result in elevated carboxyhaemoglobin levels.
* individuals subject to conditions that result in elevated levels of methaemoglobin.
* individuals with arterial cannulation or hypoxia at FiO2 = 0,21

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-12-14 (Estimated); Study Completion 2020-04-14 (Estimated)

PRIMARY OUTCOMES:
A_rms determination | Within 3 months after subject recruitment, the calibration and ARMS determination should have been performed.
  After calibration of the NightOwl SpO2 software module, the A_rms metric will be computed. This metric constitutes the performance metric proposed by ISO 80601-2-61:2011 Annex CC: Determination of accuracy. This metric captures the bias and precision of the computed SpO2 values compared to the benchmark.

CONTACTS AND LOCATIONS:
Locations (1):
- CMC, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No